CLINICAL TRIAL: NCT06252831
Title: Study of the Safety and Tolerability of the Broad-spectrum Probiotic Medicine "AS-Probionorm" Against Human Intestinal Infections in Healthy Volunteers Produced by Industrial Microbiology LLP (Phase 1)
Brief Title: Study of the Safety and Tolerability of the Broad-spectrum Probiotic Medicine "AS-Probionorm"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Industrial Microbiology LLP (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ПМ-001-23г
Record Dates: First submitted 2024-01-25; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Intestinal Infections; Dysbacteriosis
Keywords: probiotic; intestinal infections; dysbiosis; lactic acid bacteria; phase 1 of clinical trial
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Intervention Model Description: Objectives of the study: Determine the safety and tolerability of the study medicine "AS-Probionorm" (powder 1 g in a sachet) in healthy study subjects.
  The study included the following stages:
  Stage 1 of the study (introductory stage) included recruitment and screening of healthy volunteers - study participants, signing of informed consent, medical examination and laboratory tests.
  Stage 2 of the study (baseline control stage) included clinical measurements before the start of the study (baseline measurements) on each subject to obtain baseline data, which were then compared with the results after the end of the study.
  Stage 3 of the study (the stage of dynamic observation of the treatment effect and safety monitoring after the study) included clinical observations in each subject daily during the use of the study medicine and a week after the last use (21 days in total).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): 1 sachet (1 g) take 2 times a day with an interval of 12 hours. The duration of taking the medicine is 7 days. The study is carried out on an outpatient basis. The total duration of each subject's participation in the clinical trial is no more than 21±1 days.
  Interventions: Drug: "AS-Probionorm"

INTERVENTIONS:
Drug: "AS-Probionorm" — Dosage form - powder for the preparation of a solution for oral administration. Dosage regimen -1 sachet (1 g) take 2 times a day with an interval of 12 hours. Apply 15-20 minutes before meals in the morning and evening. Before use, the medicine is mixed with 30-50 ml of boiled water at room temperature, resulting in a cream-colored suspension. The resulting aqueous suspension should be drunk without achieving complete dissolution. The diluted drug cannot be stored. The duration of taking the medicine is 7 days. The study is carried out on an outpatient basis.
  The total duration of each subject's participation in the clinical trial is no more than 21 ± 1 days. Throughout the entire study period, the research subject has the opportunity to contact the research team on all questions relating to the nature of this study. After completion of the entire observation period of 21 days, there is no follow-up of study subjects under the trial protocol.

SUMMARY:
The subject of this clinical trial is the medicine "AS-Probionorm". Pharmacological group - Antidiarrheal drugs. Antidiarrheal microorganisms. Microorganisms that produce lactic acid.

The investigational probiotic medicine "AS-Probionorm" was created on the basis of an association of lactic acid bacteria with targeted action for oral use for the treatment of inflammatory and infectious diseases of the human gastrointestinal tract.

The first phase of a clinical trial is the first test of a medicine conducted on healthy volunteers to establish tolerability and safety.

According to the goal and objectives of the phase I clinical trial, the main parameter is to study the safety and tolerability of the medicine throughout the entire study period.

Phase I of the clinical trial of the medicine included 20 healthy subjects of both sexes aged 18-50 years. Clinical and laboratory parameters to characterize the safety of the medicine: medical history, physical examination, ECG, general and biochemical blood tests, urine and stool tests.

Selection and Exclusion of Subjects: Prior to inclusion in a clinical trial, each trial subject must first sign an Informed Consent Form for Participation in the Study, followed by a screening examination of each subject, including a variety of procedures, medical history, and physical examination. Each subject participating in the survey will be assigned an identification number.

Study design: open-label, single-center, phase I of clinical trial. Dosage regimen - 1 sachet (1 g) 2 times a day with an interval of 12 hours. The total duration of study subjects' participation in the study is 21 days. Tolerability of the study drug: Tolerability of the drug will be assessed based on subjective symptoms and sensations reported by patients and objective data obtained by the investigator during the study. The frequency of occurrence and nature of adverse reactions are also taken into account.

The degree of tolerability of the study drug will be determined in three gradations: intolerance, absence of undesirable drug reactions (side reactions), undesirable drug reactions (side effects) not classified as serious.

Ethical and Legal Issues in Clinical Research: This clinical trial will be conducted in accordance with the principles set forth by the 18th World Medical Assembly (Helsinki, 1964) and the ICH guidelines for good clinical practice (GCP), and in accordance with all international and national laws and regulations.

DETAILED DESCRIPTION:
Dosage form of the medicine "AS-Probionorm" (powder for the preparation of solution for oral administration) - 1 g in a sachet.

Pharmacological group - Antidiarrheal drugs. Antidiarrheal microorganisms. Microorganisms that produce lactic acid.

Introduction:

Acute intestinal infections (AII) are one of the pressing health problems in all countries. The complexity of their treatment is associated with the massive irrational use of antibiotics and chemotherapeutic drugs, which has led to the development of multidrug resistance in pathogens. Therefore, the modern strategy for the treatment of acute intestinal infections gives priority to therapeutic measures aimed at correcting intestinal microbiocenosis to eliminate the source of infection localized in the intestine.

The main idea is to conduct clinical studies of the domestic medicinal probiotic medicine "AS-Probionorm" based on the association of lactic acid bacteria of targeted action for oral use for the treatment of inflammatory and infectious diseases of the human gastrointestinal tract.

During preclinical trials, it was established that the drug exhibits high antimicrobial activity, therapeutic and prophylactic effectiveness, as well as safety during use.

The purpose of the study was to study the safety and tolerability of the study medicine "AS-Probionorm" in healthy study subjects.

Phase I of the clinical trial of the drug included 20 healthy subjects of both sexes aged 18-50 years. Clinical and laboratory parameters to characterize the safety of the drug: medical history, physical examination, ECG, general and biochemical blood tests, urine and stool tests.

Study design: open-label, single-center, phase I clinical trial. Dosage regimen: 1 sachet (1 g) 2 times a day with an interval of 12 hours. The study drug should be used 15-20 minutes before meals in the morning and evening. Before use, the medicine is mixed with 30-50 ml of boiled water at room temperature, resulting in a cream-colored suspension. The resulting water suspension should be drunk. The duration of taking is 7 days.

The study will be carried out on an outpatient basis. The total duration of study subjects' participation in the study is 21 days. On days 1, 8, 15, 21, a medical examination and laboratory tests will be carried out.

The duration of the study course of 21 days is determined by studying the possibility of developing local toxic and allergic reactions at the dosages recommended to identify the therapeutic effect.

Tolerability of the drug will be assessed based on subjective symptoms and sensations reported by patients and objective data obtained by the investigator during the study. The frequency of occurrence and nature of adverse reactions are also taken into account. The degree of tolerability of the study drug will be determined by three gradations: intolerance, absence of undesirable drug reactions (side reactions), undesirable drug reactions (side effects) not classified as serious.

Statistical analysis of data is carried out based on the results of collecting anamnestic, clinical data, as well as data from laboratory and instrumental studies. The volume of consultations, examinations and concomitant treatment carried out before the study is also recorded. Data collection will be carried out using an approved form - Individual Registration Card.

Ethical and legal issues in clinical research Ethical principles: The clinical trial will be conducted in accordance with the principles formulated by the 18th World Medical Assembly (Helsinki, 1964) and the ICH guidelines for good clinical practice (GCP).

Laws and Regulations: The clinical trial will be conducted in accordance with all international laws and guidelines, as well as national laws and regulations in accordance with any applicable guidelines.

Data collection, maintenance and storage of records. Data collection will be carried out electronically and, partially, in paper form.

The Investigator must maintain all research documentation (electronic and paper) in confidence and take steps to prevent accidental or premature destruction of this documentation.

The Investigator must retain all study documentation for a minimum of fifteen (15) years after completion or premature termination of the clinical trial.

However, if a longer period is required, applicable legal requirements must be taken into account.

The investigator must notify the sponsor before destroying any important study documents following completion or premature termination of a clinical trial.

Financing and insurance. All financing and insurance issues will be determined in the agreement concluded between the Sponsor and the Contractor.

Publications. The Investigator agrees not to publish or report the study and/or its results without the prior written permission of the study sponsor, noting that the sponsor will not withhold such permission without reasonable cause. The researcher will not use the sponsor's name in any promotional material or publication without the sponsor's prior written consent. The sponsor will not use the name of the investigator and/or his/her collaborators in promotional materials or publications without first obtaining his/their written consent. The sponsor has the right to publish the study results at any time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes aged 18-50 years with a verified state of health, absence of chronic and acute systemic and intestinal diseases; for women - a negative pregnancy test and agreement to adhere to adequate methods of contraception.
* Voluntary desire to participate in the study.

Exclusion Criteria:

* Persons with a history of allergies to milk, and during screening (drug, pollen and other types), individual hypersensitivity to the components of the drug;
* Persons with chronic diseases (tuberculosis, hepatitis, HIV infection, diabetes mellitus, cancer, blood diseases), chronic renal failure, chronic liver failure, exacerbations of chronic diseases;
* Persons taking parallel participation in clinical trials of other drugs or participating in them for 3 months from the start of the current study;
* Persons planning to participate in studies should not take any other medications for 2 weeks before clinical studies of the test drug;
* Persons from the category of "vulnerable patients" (homeless, military personnel, incapacitated, patients in emergency conditions, other persons who may be under pressure);
* Pregnancy and breastfeeding;
* The research subject does not agree to perform the procedures required by the protocol and is unable to adhere to the procedure schedule.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-02 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2023-10-14 (Actual)

PRIMARY OUTCOMES:
Safety assessment criteria | 21 days
  Absence of clinically significant changes in the parameters of general blood and urine tests, biochemical blood tests, and microbiological studies of stool of the study subjects during the study period.
Tolerability of the study drug | 21 days
  The degree of tolerability of the study drug will be determined in three gradations:
  * Intolerance - the appearance of local signs of allergy/pseudoallergy and systemic signs - tachycardia (heart rate more than 90 per minute within 30 minutes after administration), decreased blood pressure (less than 100/60 mmHg within 30 minutes after application), serious adverse drug reactions.
  * Absence of unwanted drug reactions (side reactions).
  * Adverse drug reactions (side effects) that are not classified as serious.

CONTACTS AND LOCATIONS:
Overall Officials: Ilyas Kulmagambetov, Doctor of Med. Sc., Principal Investigator — Centre for Clinical Medicine and Research LLP
Locations (1):
- MIPO Clinic LLP, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A.K. Sadanov, N.N. Gavrilova, I.A. Ratnikova, S.E. Orazymbet, E.Zh. Shorabayev, Zh.T. Musabekov, R.Zh. Kaptagay, L.E. Protasyuk, L.A. Kosheleva, S.B. Dzhailyauova Association of bacteria for the production of a medicinal probiotic preparation with a wide spectrum of antimicrobial action // Microbiology and virology. - ISSN 2304-585X. - No. 1 (40) 2023. -- pp. 116-126. - doi: 10.53729/MV-AS.2023.01.07; IF-0.038.
- [Background] Sadanov A.K., Gavrilova N.N., Ratnikova I.A., Orazymbet S.E., Shorabayev E.Zh., Protasyuk L.E. Antimicrobial activity of the therapeutic and prophylactic probiotic drug "AS-Probionorm" // Proc. on Sat. mater. Intl. scientific-practical conf. "Biotechnology and biological safety: achievements and development prospects", dedicated to the 65th anniversary of the Research Institute for Biological Safety Problems. - Almaty. - September 6-8, 2023 - P. 134. - UDC 57/60 BBK 28/30.16 B63. ISBN 978-601-305-533-6.
- [Background] A.K. Sadanov, N.N. Gavrilova, I.A. Ratnikova, S.E. Orazymbet, L.E. Protasiuk, A.D. Massirbaeva Technology for the production of Lyophilizate of an association of Lactic acid bacteria included in the Medicinal product AS-Probionorm // Research J. Pharm. and Tech. 16(11):5334-5340. - November 2023. - DOI: 10.52711/0974-360X.2023.00864. - ISSN 0974-3618 (Print), 0974-360X (Online). Q2, 56th percentile.